CLINICAL TRIAL: NCT03450499
Title: Analgesia Effects of Intravenous Ketamine After Spinal Anesthesia for Non-elective Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, prahlad adhikari, doctor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRC/1089/017
Record Dates: First submitted 2018-02-18; First posted 2018-03-01 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Non Elective Cesarean Section and Ketamine Analgesia
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- analgesic effects of ketamine (Experimental): the experimental group will receive ketamine intravenously at 0.25 mg per kg before skin incision.
  Interventions: Drug: Ketamine
- placebo (Placebo Comparator): they will receive same volume of 0.9% normal saline as calculated for experimental group before skin incision.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — the analgesic affects of ketamine will be compared between the experimental and placebo group.
  Other Names: ketamine hydrochloride
  Arms: analgesic effects of ketamine
Drug: Placebo — the analgesic requirement will be calculated in placebo group.
  Arms: placebo

SUMMARY:
This randomized double blind study will be conducted in pregnant woman planned for non elective cesarean section under spinal anesthesia. Ketamine group will receive intravenous 0.25 mg/kg and placebo group will receive same amount of normal saline after spinal anesthesia prior to skin incision. Postoperative outcomes measures are total opioid consumption and pain scores for 24 hrs.

ELIGIBILITY:
Inclusion Criteria:

* • All women at term(>or =37 weeks of gestation)

  * Healthy
  * American Society of Anesthesiologists(ASA) class1 and 2
  * Women undergoing non-elective caesarean section whose anesthetic plan is for spinal anesthesia with bupivacaine and fentanyl

Exclusion Criteria:

* • Women with American society of anesthesiologist physical status>2

  * Body mass index >or =40 kg per square meter
  * Height <150 cm
  * Any contraindication to the spinal anesthesia
  * History of substance abuse
  * History of hallucinations
  * Chronic opioid therapy
  * Chronic pain or on any pain medication currently
  * Patient with maternal complications,like cardiovascular disease pre-eclampsia,diabetes,multiple gestation,known fetal abnormality
  * Cases with severely compromised fetus where immediate administration of general anesthesia is required.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Total opioid requirement postoperatively | 24 hrs
  Total opioid required up to 24 postoperatively in ketamine and placebo group.

SECONDARY OUTCOMES:
Postoperative numerator rating scores(NRS)up to 24 hrs . postoperative ) | 24 hrs
  • Postoperative NRS Scores (on arrival to Post operative care unit), 2, 4, 6, 8, 12 and 24 h ).The NRS ranges from 0- 10 and 0 refers to no pain and 10 means extreme possible pain perceived.
Time to first perception of pain | 24 hrs
  Time to first perception of pain
Incidence of side effects | 24 hrs
  Incidence of post operative nausea and vomiting, shivering, sedation scores, side effects related to ketamine during the first 24h

CONTACTS AND LOCATIONS:
Locations (1):
- BP Koirala Institute of Health Sciences (BPKIHS), Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adhikari P, Subedi A, Sah BP, Pokharel K. Analgesic effects of intravenous ketamine after spinal anaesthesia for non-elective caesarean delivery: a randomised controlled trial. BMJ Open. 2021 Jun 30;11(6):e044168. doi: 10.1136/bmjopen-2020-044168. PMID 34193480